CLINICAL TRIAL: NCT06918834
Title: Efficacy of Immediate Allogeneic Hematopoietic Stem Cell Transplantation Versus Bridging Therapy Followed by Transplantation in Higher-Risk Myelodysplastic Syndrome Patients: A Multicenter, Randomized Controlled, Open-Label, Phase 2 Clinical Trial
Brief Title: Efficacy of Immediate Allogeneic Hematopoietic Stem Cell Transplantation Versus Bridging Therapy Followed by Transplantation in Higher-Risk Myelodysplastic Syndrome Patients
Acronym: ImmBridge
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025016
Record Dates: First submitted 2025-03-11; First posted 2025-04-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate HSCT Group (Experimental)
  Interventions: Other: Immediate HSCT Group
- Bridging Therapy Group (Active Comparator)
  Interventions: Other: Bridging Therapy Group

INTERVENTIONS:
Other: Immediate HSCT Group — Patients undergo direct allogeneic HSCT.
  Arms: Immediate HSCT Group
Other: Bridging Therapy Group — Patients receive one to two cycles of bridging therapy before undergoing allogeneic HSCT.
  o Bridging Therapy Regimen: Hypomethylating agents (HMA) alone or HMA-based combination chemotherapy, e.g., azacitidine (AZA) 100 mg/day + venetoclax (VEN) 400 mg/day for 7 days. Targeted therapies (e.g., IDH1 inhibitors) will be used for eligible patients.
  Arms: Bridging Therapy Group

SUMMARY:
This study aims to evaluate whether immediate allogeneic hematopoietic stem cell transplantation (HSCT) is non-inferior to HSCT following bridging therapy in patients with higher-risk myelodysplastic syndrome (HR-MDS).

DETAILED DESCRIPTION:
A total of 236 patients will be randomized in a 1:1 ratio into the immediate transplantation group (n=118) and the disease control group (n=118). The study will continue until at least 124 events occur.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. High relapse risk MDS, defined by:

   * IPSS-R score ≥3.5.
   * IPSS-M stratification as intermediate-high, high, or very high risk.
3. Eligible for allogeneic HSCT (including matched or mismatched related/unrelated donor transplantations).
4. Karnofsky Performance Status (KPS) ≥60.
5. Signed informed consent.

Exclusion Criteria:

1. Severe organ dysfunction:

   * Left ventricular ejection fraction <50%.
   * Oxygen supplementation requirement.
   * Serum bilirubin >1.5x upper limit of normal (unless due to Gilbert syndrome) or AST/ALT >5x upper limit of normal.
   * Estimated glomerular filtration rate (eGFR) <50 mL/min.
2. History of prior allogeneic HSCT.
3. Any condition deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
2-year Disease-Free Survival (DFS) post-HSCT | 2-year
  Defined as the time from transplantation to two years post-HSCT, with primary events including death or failure to achieve CR or CR equivalent at the time of assessment

SECONDARY OUTCOMES:
Cumulative Incidence of Allogeneic HSCT | The proportion of patients who undergo HSCT at 4, 8, 16, and 24 weeks post-randomization.
  The proportion of patients who undergo HSCT at 4, 8, 16, and 24 weeks post-randomization.
Complete Remission (CR) or CR Equivalent Rate from Randomization | 2-year
  The percentage of patients achieving CR or CR equivalent, defined as the first documented occurrence.
2-year Overall Survival (OS) post-HSCT | 2-year
  Defined as the time from HSCT to death from any cause within two years.
2-year Leukemia-Free Survival (LFS) from Randomization | 2-year
  The time from randomization to the occurrence of disease progression, relapse, or death from any cause within two years.
2-year Quality of Life (QoL) Assessment: 2-year Quality of Life (QoL) Assessment from Randomization | 2-year
  Defined as the assessment of patient-reported QoL starting from randomization over a 2-year period, evaluated using the EORTC QLQ-C30 questionnaire.
Molecular Clearance Rate | 2-year
  Molecular clearance was defined by two consecutive blood samples obtained at least 4 weeks apart after that were negative for driver mutations in a patient who had been positive before transplantation.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University People's Hospital, Beijin, Beijing Municipality
  - Zhengzhou University First Affiliated Hospital, Zhengzhou, Henan
  - The 960th Hospital of the Joint Service Support Force of the Chinese People's Liberation Army, Jinan, Shandong
  - People's Liberation Army The General Hospital of Western Theater Command, Chengdu, Sichuan
  - The Second Hospital of Hebei Medical University, Shijia Zhuang

IPD SHARING:
Plan to Share IPD: No